CLINICAL TRIAL: NCT00476099
Title: A 48-week, Double Blind, Double Dummy, Randomised, Multinational, Multicentre, 3-arm Parallel Group Clinical Study of "Fixed Combination" Beclometasone Dipropionate Plus Formoterol Fumarate Administered Via pMDI With HFA-134a Propellant Versus "Fixed Combination" Budesonide Plus Formoterol DPI Versus Formoterol DPI in Patients With Stable Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Efficacy and Safety Study of Beclometasone/Formoterol Single Inhaler in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DM/PR/033011/005/05; 2006-002489-20 (EudraCT Number)
Record Dates: First submitted 2007-05-18; First posted 2007-05-21 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone; Formoterol Fumarate; Budesonide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) pMDI (Experimental)
  Interventions: Drug: Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) pMDI; Drug: Budesonide 200 µg plus formoterol 6 µg DPI; Drug: Formoterol 12 µg DPI
- Budesonide 200 µg plus formoterol 6 µg DPI (Active Comparator)
  Interventions: Drug: Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) pMDI; Drug: Budesonide 200 µg plus formoterol 6 µg DPI; Drug: Formoterol 12 µg DPI
- Formoterol 12 µg DPI (Active Comparator)
  Interventions: Drug: Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) pMDI; Drug: Budesonide 200 µg plus formoterol 6 µg DPI; Drug: Formoterol 12 µg DPI

INTERVENTIONS:
Drug: Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) pMDI — Beclomethasone 100 µg plus formoterol 6 µg (CHF1535) two puffs via oral inhalation twice a day at 8.00 a.m. and 8.00 p.m.
Drug: Budesonide 200 µg plus formoterol 6 µg DPI — two oral inhalations twice a day at 8.00 a.m. and 8.00 p.m.
Drug: Formoterol 12 µg DPI — one oral inhalation twice a day at 8.00 a.m. and 8.00 p.m.

SUMMARY:
To evaluate the 1-year efficacy and safety of the fixed combination beclometasone/formoterol pMDI in a twice daily regimen in patients with stable severe COPD.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the long-term efficacy and safety of the fixed combination beclometasone/formoterol pMDI in a twice daily regimen in patients with stable severe COPD. Patients are randomised to receive either beclometasone/formoterol or budesonide/formoterol DPI or formoterol DPI during 48 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD (according to GOLD guidelines)
* FEV1 > or equal 30% and < 50% of predicted normal post-bronchodilator (and at least 0.7 L absolute value)
* COPD symptoms for at least 2 years
* At least 1 exacerbation requiring medical intervention (oral corticosteroid and/or antibiotic treatment and/or need for a visit to an emergency department and/or hospitalization) within 2-12 months before screening
* Current or previous smoker with a cumulative exposure to smoke of more than 20-pack year

Exclusion Criteria:

* Current or past diagnosis of asthma, or any evidence suggestive of asthma
* Positive FEV1 reversibility test
* Clinically significant or unstable concurrent diseases, including clinically significant laboratory abnormalities
* Acute COPD exacerbation or lower tract infection and/or treatment with oral or injectable corticosteroids and antibiotics in the 2 months before screening or during run-in
* Long term oxygen therapy

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 828 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Number of COPD exacerbations and pre-dose morning FEV1 | one year treatment

SECONDARY OUTCOMES:
Other pulmonary function parameters, | one year treatment
COPD symptom scores and Quality of Life, | one year treatment
safety and tolerability | one year treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter M.A. Calverley, Professor, Principal Investigator — Department of Medicine, Clinical Sciences Center University Hospital Aintree, Liverpool, United Kingdom
Locations (1):
- Thomas Similowski, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Chiesi commits to sharing with qualified scientific and medical Researchers, conducting legitimate research, Patient-level Data, Study-level Data, the Clinical Protocol and the full CSR, providing access to clinical trial information consistently with the principle of safeguarding commercially confidential information and patient privacy. Any shared Patient-level Data is anonymized to protect personally identifiable information.
  Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
Access Criteria: Chiesi access criteria and complete process for clinical data sharing is available on the Chiesi Group website.
URL: https://www.chiesi.com/en/chiesi-clinical-trial-data-request-portal/

REFERENCES:
- [Background] Singh D, Corradi M, Spinola M, Petruzzelli S, Papi A. Extrafine beclometasone diproprionate/formoterol fumarate: a review of its effects in chronic obstructive pulmonary disease. NPJ Prim Care Respir Med. 2016 Jun 16;26:16030. doi: 10.1038/npjpcrm.2016.30. PMID 27309985
- [Result] Calverley PM, Kuna P, Monso E, Costantini M, Petruzzelli S, Sergio F, Varoli G, Papi A, Brusasco V. Beclomethasone/formoterol in the management of COPD: a randomised controlled trial. Respir Med. 2010 Dec;104(12):1858-68. doi: 10.1016/j.rmed.2010.09.008. Epub 2010 Oct 20. PMID 20965712
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=2006-002489-20
- See also: CSR Synopsis available in the CHIESI Clinical Study Register — https://www.chiesi.com/clinic/82_CSR_Synopsis_DM-PR-033011-005-05.pdf